CLINICAL TRIAL: NCT05663749
Title: Efficacy and Safety of Add-on Topiramate vs Metformin on Cardio-Metabolic Profile in Patients With Schizophrenia on Atypical Antipsychotics With Metabolic Syndrome: a Randomized Controlled Trial
Brief Title: Topiramate vs Metformin on Cardio-Metabolic Profile in Schizophrenia on Atypical Antipsychotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, BISWA RANJAN MISHRA, Additional Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIIMS BBSR/PG Thesis/2021-22
Record Dates: First submitted 2021-12-04; First posted 2022-12-23 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2022-12

CONDITIONS: Metabolic Syndrome; Schizophrenia
Keywords: Metabolic Syndrome; Schizophrenia; Atypical antipsychotics; Topiramate; Metformin
MeSH Terms: conditions — Metabolic Syndrome; Schizophrenia | interventions — Metformin; Topiramate; Topaz resin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin arm (Active Comparator): 1000mg for 8 weeks
  Interventions: Drug: Metformin
- Topiramate arm (Experimental): 50mg for 8 weeks
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Metformin — 1000mg for 8 weeks
  Other Names: Dibeta SR; Metgen; Glycomet
  Arms: Metformin arm
Drug: Topiramate — 50mg for 8 weeks
  Other Names: Topamax; Topirol; Topaz
  Arms: Topiramate arm

SUMMARY:
Metabolic syndrome is common in patients of schizophrenia. It can add to morbidity, loss of functionality and discontinuation of antipsychotic medication. Apart from metformin, there are limited treatment options as add on-s to antipsychotics for treatment of metabolic syndrome. There have been placebo-controlled studies of Topiramate as an adjuvant but the present study would be the first head-on trial between these drugs for treatment of metabolic syndrome in patients of schizophrenia.

If the outcome measures show a significant improvement with add on topiramate when compared with Metformin, then add on Topiramate can be a preferred treatment for metabolic syndrome in patients with schizophrenia on atypical antipsychotics. The adverse effects of Metformin can be side-stepped and Topiramate can also be given in conditions which are contraindications for Metformin. Thus, Topiramate can be a good alternative to metformin especially in conditions like liver, cardiac and renal impairment where metformin use should be avoided. Topiramate can not only improve metabolic parameters but can also have a beneficial effect on the symptom severity of schizophrenia. Thus, it can be a good augmentation drug to be used along with antipsychotics in these patients.

DETAILED DESCRIPTION:
Study Design: The proposed study will be a randomised, parallel arm, active controlled, open label, clinical trial.

Study Setting: The proposed study will be conducted at the out-patient (OP) and the in-patient (IP) settings of the Department of Psychiatry, All India Institute of Medical Sciences, Bhubaneswar.

Study Groups: The study population will comprise of 60 patients with schizophrenia (F20 according to ICD 10 DCR) on atypical antipsychotics for more than 3 months diagnosed with metabolic syndrome.

Sample size: Sample size calculation has been done based on the expected difference in the cardiovascular risk scoring (QRISK3), the primary outcome measure of our study. Sample size of 23 per group will achieve a power of 80%, to detect the difference of 5% in cardiovascular risk scoring (QRISK3) between the groups with standard deviation as 6.0 and a level of significance 0.05. Assuming an attrition rate of 25%, 30 patients will be recruited per group.

Details of Control(s): It is an active controlled study where the control group will receive add-on metformin along with the ongoing atypical antipsychotic.

Details of intervention:

The patients who are randomized to Topiramate group will be receiving Topiramate at a stable dose of 50 mg/day during the study period that is for 8 weeks along with the ongoing atypical antipsychotic.

The patients who are randomized to Metformin group will be receiving Metformin at dose of 500 mg/day twice a day, a total of 1000 mg/day for 8 weeks along with the ongoing atypical antipsychotic.

Duration of study: The study will be conducted for a period of 18 months

Investigation specifically related to Protocols:

The following Psychiatric scales will be used:

1. PANSS: The Positive and Negative Syndrome Scale
2. CGI-SCH Scales: The Clinical Global Impression-Schizophrenia scale (for Severity and Improvement) The following investigations will be done for cardio-metabolic profile;

a) QRISK3 b) Lipid profile c)Fasting serum insulin by ELISA for insulin resistance (HOMA-IR) d)Fasting blood glucose for insulin resistance (HOMA-IR)

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with schizophrenia (F20 according to ICD-10 DCR) on a stable dose of atypical antipsychotic for more than 3 months.
* Patients with metabolic syndrome (as per NCEP ATP III Definition).
* Patients above 25 years of age of either gender.
* Legally authorized representative (LAR) giving voluntary written consent for participation in the study.

Exclusion Criteria:

* Patients on combination of antipsychotics.
* Patients having any contraindication for Metformin/Topiramate.
* History of any psychoactive substance use in harmful use or dependence pattern except tobacco.
* Any co-morbid medical, psychiatric or neurological disorders like hypertension, coronary artery disease, hypothyroidism, arthritis.
* History of any significant head injury or organic diseases.
* Pregnant and breastfeeding females.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Change in the QRISK3 score. | 8 weeks
  QRISK3 (QRESEARCH cardiovascular risk algorithm)2018 algorithm- used for calculating the cardiovascular risk in the upcoming 10 years. It is measured for the age group of 25 to 84 years using information like age, weight, height, BMI, Lipid profile, past history of CKD, angina, migraine etc. Higher score indicates higher risk.

SECONDARY OUTCOMES:
Change in the LDL/HDL ratio(Low density lipoprotein/High density lipoprotein).Higher ratio indicates higher risk | 8 weeks
  Calculated from the lipid profile
Change in Insulin Resistance (HOMA-IR)(homeostasis model assessment-estimated insulin resistance ). | 8 weeks
  Calculated from serum insulin level and fasting glucose level according to the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Change in Positive and negative syndrome scale | 8 weeks
  Positive and negative syndrome scale, a scale used to measure the symptom severity in patients of schizophrenia including positive, negative and general psychopathology.Higher scores indicate more severity of illness.Maximum score 30 and maximum 210
Change in Clinical Global Impression-Schizophrenia scale | 8 weeks
  Scale that is used to measure the baseline severity, change in severity of illness with treatment and global improvement. More score indicates more impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Biswa Ranjan Mishra, MD, DPM, Principal Investigator — All India Institute of Medical Sciences, Bhubaneswar
Locations (1):
- Dept of Psychiatry, Aiims, Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saha S, Chant D, McGrath J. A systematic review of mortality in schizophrenia: is the differential mortality gap worsening over time? Arch Gen Psychiatry. 2007 Oct;64(10):1123-31. doi: 10.1001/archpsyc.64.10.1123. PMID 17909124
- [Background] DE Hert M, Schreurs V, Vancampfort D, VAN Winkel R. Metabolic syndrome in people with schizophrenia: a review. World Psychiatry. 2009 Feb;8(1):15-22. doi: 10.1002/j.2051-5545.2009.tb00199.x. PMID 19293950
- [Background] Rummel-Kluge C, Komossa K, Schwarz S, Hunger H, Schmid F, Lobos CA, Kissling W, Davis JM, Leucht S. Head-to-head comparisons of metabolic side effects of second generation antipsychotics in the treatment of schizophrenia: a systematic review and meta-analysis. Schizophr Res. 2010 Nov;123(2-3):225-33. doi: 10.1016/j.schres.2010.07.012. Epub 2010 Aug 7. PMID 20692814
- [Background] Zheng W, Li XB, Tang YL, Xiang YQ, Wang CY, de Leon J. Metformin for Weight Gain and Metabolic Abnormalities Associated With Antipsychotic Treatment: Meta-Analysis of Randomized Placebo-Controlled Trials. J Clin Psychopharmacol. 2015 Oct;35(5):499-509. doi: 10.1097/JCP.0000000000000392. PMID 26280837
- [Background] Flory J, Lipska K. Metformin in 2019. JAMA. 2019 May 21;321(19):1926-1927. doi: 10.1001/jama.2019.3805. PMID 31009043
- [Background] Goh KK, Chen CH, Lu ML. Topiramate mitigates weight gain in antipsychotic-treated patients with schizophrenia: meta-analysis of randomised controlled trials. Int J Psychiatry Clin Pract. 2019 Mar;23(1):14-32. doi: 10.1080/13651501.2018.1449864. Epub 2018 Mar 20. PMID 29557263
- [Background] Lawrence D, Hancock KJ, Kisely S. The gap in life expectancy from preventable physical illness in psychiatric patients in Western Australia: retrospective analysis of population based registers. BMJ. 2013 May 21;346:f2539. doi: 10.1136/bmj.f2539. PMID 23694688
- [Background] Allison DB, Mentore JL, Heo M, Chandler LP, Cappelleri JC, Infante MC, Weiden PJ. Antipsychotic-induced weight gain: a comprehensive research synthesis. Am J Psychiatry. 1999 Nov;156(11):1686-96. doi: 10.1176/ajp.156.11.1686. PMID 10553730
- [Background] Praharaj SK, Jana AK, Goyal N, Sinha VK. Metformin for olanzapine-induced weight gain: a systematic review and meta-analysis. Br J Clin Pharmacol. 2011 Mar;71(3):377-82. doi: 10.1111/j.1365-2125.2010.03783.x. PMID 21284696
- [Background] Chen CH, Chiu CC, Huang MC, Wu TH, Liu HC, Lu ML. Metformin for metabolic dysregulation in schizophrenic patients treated with olanzapine. Prog Neuropsychopharmacol Biol Psychiatry. 2008 May 15;32(4):925-31. doi: 10.1016/j.pnpbp.2007.11.013. Epub 2007 Nov 17. PMID 18082302
- [Background] de Silva VA, Suraweera C, Ratnatunga SS, Dayabandara M, Wanniarachchi N, Hanwella R. Metformin in prevention and treatment of antipsychotic induced weight gain: a systematic review and meta-analysis. BMC Psychiatry. 2016 Oct 3;16(1):341. doi: 10.1186/s12888-016-1049-5. PMID 27716110
- [Background] Narula PK, Rehan HS, Unni KE, Gupta N. Topiramate for prevention of olanzapine associated weight gain and metabolic dysfunction in schizophrenia: a double-blind, placebo-controlled trial. Schizophr Res. 2010 May;118(1-3):218-23. doi: 10.1016/j.schres.2010.02.001. Epub 2010 Mar 7. PMID 20207521
- [Background] Egger C, Muehlbacher M, Schatz M, Nickel M. Influence of topiramate on olanzapine-related weight gain in women: an 18-month follow-up observation. J Clin Psychopharmacol. 2007 Oct;27(5):475-8. doi: 10.1097/jcp.0b013e31814b98e5. PMID 17873679
- [Background] Ellinger LK, Ipema HJ, Stachnik JM. Efficacy of metformin and topiramate in prevention and treatment of second-generation antipsychotic-induced weight gain. Ann Pharmacother. 2010 Apr;44(4):668-79. doi: 10.1345/aph.1M550. Epub 2010 Mar 16. PMID 20233913
- [Background] Ince B, Altinbas K. [Ten-Year Risk of Cardiovascular Disease in Patients with Bipolar Disorder]. Turk Psikiyatri Derg. 2020 Winter;31(4):225-231. doi: 10.5080/u25270. Turkish. PMID 33454933
- [Background] Tang Q, Li X, Song P, Xu L. Optimal cut-off values for the homeostasis model assessment of insulin resistance (HOMA-IR) and pre-diabetes screening: Developments in research and prospects for the future. Drug Discov Ther. 2015 Dec;9(6):380-5. doi: 10.5582/ddt.2015.01207. PMID 26781921
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518